CLINICAL TRIAL: NCT06796894
Title: Comparison of Symptoms, Respiratory Dysfunction and Frailty Level in Allergic and Eosonophilic Asthmatics
Brief Title: Symptoms, Respiratory Dysfunction and Frailty Level in Allergic and Eosonophilic Asthmatics
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, Professor, Hacettepe University
Other Study IDs: SBA 24/477
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Asthma; Respiratory Disease; Fragility
Keywords: Asthma; Respiratory Dysfunction; Fragility
MeSH Terms: conditions — Asthma; Respiration Disorders; Dyspnea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to determine the level of respiratory dysfunction, symptoms and frailty in patients with asthma according to different endophenotypes (allergic and eosonophilic asthma). In the light of the data obtained, it is thought that rehabilitation approaches that can be determined according to different endophenotypes in line with the evaluated parameters will guide health professionals working in this field.

Hypotheses H0: There is no difference between allergic and eosonophilic asthmatics in terms of pulmonary function, respiratory dysfunction, symptoms, dyspnoea, fatigue, rhinitis, perception of breathlessness in activities of daily living, asthma control, level of frailty or quality of life.

H1: There is a difference between individuals with allergic and eosonophilic asthma in terms of pulmonary function, respiratory dysfunction, symptoms, dyspnoea, fatigue, rhinitis, perception of breathlessness in activities of daily living, asthma control, level of frailty or quality of life.

DETAILED DESCRIPTION:
Asthma, which is characterised by variable airway obstruction and bronchial sensitivity, is an increasingly common chronic respiratory disease both globally and in our country. It is known that asthma has many phenotypes and endotypes according to its pathophysiology and some biomarkers as well as symptoms are used to determine these. The main phenotypes are allergic asthma, non-allergic asthma, late-onset asthma and asthma with permanent airflow limitation. Allergic asthma is generally defined as asthma associated with sensitisation to aeroallergens. Sensitisation to aeroallergens contributes significantly to asthma symptoms and airway inflammation. Allergic asthma is the most common asthma phenotype. It is estimated that 80% of childhood asthma and more than 50% of adult asthma cases may have an allergic component. Allergic asthma is often accompanied by a history of eczema and allergic rhinitis. Numerous biomarkers have been established to identify patients with allergic asthma, including atopy tests such as total IgE and specific IgE and skin tests for allergens.

Although allergic asthma and eosonophilic asthma have similar inflammatory processes, some differences in their definitions have been emphasised in recent studies. Type-2 inflammatory processes play a role in both endophenotypes. Current guidelines provide separate treatment recommendations for allergic and eosinophilic asthma and emphasise the need for studies to guide the clinically meaningful interpretation of asthma endophenotypes.

Asthmatic patients frequently complain of symptoms such as dyspnoea, cough and chest tightness. In addition, it is recommended that patients should be evaluated for fatigue and rhinitis. Depending on the severity of the disease, respiratory function is impaired. According to the severity of symptoms, attack status and pulmonary functions, it is determined which step of treatment to start in the newly diagnosed patient and whether asthma is under control in the patient receiving treatment. Treatment and rehabilitation approaches applied to individuals vary according to the severity and control status of asthma.

In the light of this information, it is aimed to determine the level of respiratory dysfunction, symptoms and frailty in asthmatic patients according to different endophenotypes (allergic and eosonophilic asthma). In the light of the data obtained, it is thought that rehabilitation approaches that can be determined according to different endophenotypes in line with the evaluated parameters will guide health professionals working in this field.

Demographic Information: Age, height (cm), weight (kg), gender, body mass index (kg/m2), occupation, time of asthma diagnosis and duration of the disease, curriculum vitae, family history, smoking history (pack*year), medications used will be recorded in the demographic information form.

Pulmonary Function Test: A pulmonary function test will be performed to assess the pulmonary function of individuals. Measurements will be performed based on the guidelines published by the American Respiratory Society (ATS) and the European Respiratory Society (ERS). The tests will be performed using a Spirodoc spirometer (Medical International Research, Rome, Italy). Individuals will be tested in an upright sitting position with a supported back. Before starting the test, individuals will be fitted with a nose clip and asked to grasp the mouthpiece tightly. Individuals will first be asked to inhale and exhale at tidal volume, followed by a verbal command to take a deep inspiration. Then, following the deep inspiration, they will be instructed to perform a long and rapid expiration for at least six seconds. The test will then be completed with a deep inspiration Modified Medical Research Council (mMRC) Dyspnoea Scale: Modified Medical Research Council (mMRC) Dyspnoea Scale will be used to evaluate the dyspnoea level in the study. This scale is a 5-item scale used to evaluate the relationship between dyspnoea severity and activity limitation. This scale includes five statements that determine the level of dyspnoea and patients will be asked to tick one of these statements.

Laboratory Results: Eosonophil count and Ig values will be recorded from the routine laboratory results of the patients.

Asthma Control: In the study, Asthma Control Test (ACT) will be used to assess asthma control in asthmatic individuals. The scale was developed by Nathan et al. (2004), and its validity and reliability was performed by Schatz et al. The scale, whose Turkish validity and reliability was performed by Uysal et al. (2013), is a five-point Likert-type scale and is evaluated by summing the scores. There are five statements in this scale. Patients will be asked to tick one of the appropriate 0-5 points from each statement. The maximum score of this test is 25 and the minimum score is 5. When scoring the ECT, 25 points is considered as "full control", 20-24 points as "good control" and less than 19 points as "no control". The highest score indicates the best control; scores of 19 and below indicate that the disease is not under control and that changes in treatment are required to achieve control.

COPD and Asthma Fatigue Scale: In the study, fatigue will be assessed with the COPD and Asthma Fatigue Scale. It was developed by Revicki et al. in 2010. Turkish validity and reliability was performed by Arslan and Öztunç (2013). The scale consists of 12 items graded on a 5-point Likert scale. Asthmatic individuals will be asked to tick the appropriate answer to 12 items. The total raw score of the scale is converted into a total scale score between 0-100 by summing each item score. The scale score is calculated with the formula [(Total Raw Score-12 /48) x100]. An increase in the scale score indicates an increase in the level of fatigue Nijmegen Questionnaire: Nijmegen Questionnaire will be used to evaluate respiratory dysfunction and symptoms in the study. Turkish validity and reliability was performed by Çakmak et al. (2023). The questionnaire includes 15 respiratory dysfunction and symptoms such as chest pain, feeling of tension, blurred vision, shortness of breath. Patients will be asked to tick the number (0: never, 4 very often) that best represents these symptoms. A total score will be calculated.

Control test for asthma and allergic rhinitis (CARAT): In the study, the control test for asthma and allergic rhinitis (CARAT) will be used to determine the control status of these two diseases for patients with asthma and concurrent allergic rhinitis diagnoses. The Turkish validity and reliability of the CARAT scale was performed by Öngel and Gemicioğlu (2020). CARAT is a scale consisting of 10 questions questioning upper and lower respiratory tract symptoms, effects on sleep, activity restriction and medication use in a 4-week period. For each of the questions, patients will be asked to choose one of 4 response options ranging from 0 to 3. 0 points indicates minimum control and 30 points indicates maximum control. Scoring is based on 3 parameters: total score, upper airway score (CARAT-usy) and lower airway score (CARAT-asy). Accordingly, a total score (CARAT-t) of more than 24 points, CARAT-usy of more than 8 points and CARAT-asy of 16 points or more indicate disease control.

London Chest Activities of Daily Living Scale: In the study, activities of daily living (ADL) performance will be evaluated with the London Chest ADL Scale (LCADAS). This scale was developed by Garrod et al. The Turkish validity and reliability study was conducted by Saka et al. The scale consists of 15 items in total. It includes four sub-headings: personal care (4 items), housework (6 items), physical activity (2 items) and leisure time (3 items). Individuals will be asked to give a score ranging from 0 to 5 for each item. A higher score indicates more impairment. The scale also includes a single question to determine the perception of general dyspnoea. This question will rate the degree to which the degree of dyspnoea affects the GAD on a scale of 'a lot, a little, not at all'. The total score ranges from 0-75.

FRAIL Scale: In the study, frailty will be assessed with the FRAIL scale, the reliability and validity of which was performed by Hymabaccus (2017). The FRAIL scale consists of 5 items including fatigue status, endurance, mobility, weight loss and existing diseases. The patient's fatigue status, endurance, mobility, weight loss and other diseases will be questioned and scored as 0 or 1 point according to their answer. According to the total score: 0 points is considered vigorous-not frail (non-frail), 1-2 points: pre-frail (pre-frail) and total score above 2 points: frail (frail).

Asthma Quality of Life Questionnaire (AQLQ): Asthma Quality of Life Questionnaire (AQLQ) will be used for disease-specific quality of life assessment. Turkish adaptation of the AQLQ developed by Juniper et al. will be used. The scale consists of 4 subsections with 12 questions about symptoms, 11 questions about activities, 5 questions about emotional state and 4 questions about environmental factors. For each question, the patients will be asked to give a score between 1 and 7 points (1: more limitation, 7: no limitation) for the limitations experienced due to asthma in the activities performed during the last two weeks. Calculations will be made for the total score and subsections.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35-75 years,
* Diagnosed with allergic or eosonophilic asthma according to the Global Strategy for the Prevention and Treatment of Asthma (GINA).

Exclusion Criteria:

* Known cognitive impairment,
* Having had an acute asthma attack in the last 6 weeks,
* Having changed medication in the last 4 weeks.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hacettepe University Faculty of Medicine Department of Paediatrics Patients aged 35-75 years who have been diagnosed with asthma in the Allergy and Asthma Unit and who volunteered to participate in the study will be included in the study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory Symptoms | One day
  The Nijmegen Questionnaire. The Nijmegen Questionnaire (NQ) gives a broad view of symptoms associated with dysfunctional breathing patterns. The NQ consists of 16 items to be answered on a five-point scale ranging from 'never' counted as zero to 'very often' counted as 4. The total score ranges from 0-64.

SECONDARY OUTCOMES:
Pulmonary functions | One day
  Pulmonary function testing by spirometer
Dyspnea during daily life | One day
  Modified Medical Research Council dyspnea scale: The mMRC (Modified Medical Research Council) Dyspnoea Scale is used to assess the degree of baseline functional disability due to dyspnoea.The mMRC breathlessness scale ranges from grade 0 to 4.
Asthma Control Level | One day
  Asthma Control Test: ACT assesses the frequency of shortness of breath and general asthma symptoms, use of rescue medications, the effect of asthma on daily functioning, and overall self-assessment of asthma control. The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
Fatigue level | One day
  COPD and Asthma Fatigue Scale: The scale consists of 12 items graded on a 5-point Likert type. Asthmatic individuals will be asked to mark the appropriate answer for 12 items. The total raw score of the scale is converted into a total scale score between 0-100 by adding each item score. An increase in the scale score indicates an increase in the level of fatigue
Asthma and allergic rhinit symptoms | One day
  Control of Allergic Rhinitis and Asthma Test: The CARAT questionnaire is composed of 10 questions that address upper and lower airway symptoms, sleep interference, activity limitation, and the need to increase medication over a four-week period The answers are rated on a four-point scale, with a total possible score ranging from 0 (minimum control) to 30 (maximum control).
Activities of daily living | One day
  London Chest ADL Scale: The LCADL is a standardized questionnaire to assess dyspnea resulting from ADL in COPD patients. It consists of a total of 15 items within four domains: personal care (four items), domestic (six items), physical (two items), and leisure (three items). Each item is graded from 0 to 5 with higher scores indicating more difficulty in performing ADL. The scale can be evaluated as the total score, domain scores, and item scores. There is also a single question that assesses to what degree dyspnea perception affects daily life in general. This item is answered by selecting one of following three responses: "a lot," "a little," or "not at all"
Frailty | One day
  FRAIL Scale: The 5-item FRAIL scale is scored 0 or 1 according to the answer given by the patients, and a total of 0 points is considered vigorous (non-frail), 1-2 points is considered pre-frail and >2 points is considered frail. A total score of 3 or more is considered as indicative of frailty, a score of 1 or 2 is considered indicative of prefrailty, and a score of 0 is considered as indicating resilience
Disease spesific quality of life | One day
  Asthma Quality of Life Questionnaire: It includes Symptoms (11 items), Activity Limitation (12 items, 5 of which are individualized), Emotional Function (5 items), and Environmental Exposure (4 items). Scores range 1-7, with higher scores indicating better quality of life
Laboratory testing | One day
  The levels of eosinophil and Ig will be recorded from medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Calik Kutukcu, Principal Investigator — Hacettepe University; Aynur Demirel, PhD, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided